CLINICAL TRIAL: NCT05250765
Title: Comparison of Efficiency and Effectiveness of Two Types of Bonded Orthodontic Retainers: an RCT.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-08508
Record Dates: First submitted 2022-01-11; First posted 2022-02-22 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Relapse
Keywords: Orthodontic retainers; Isolation; Bonding; Twistflex retainer; Coaxial retainer; OrthoflexTech retainer; Fixed retainer
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Intervention Model Description: 4 study groups are possible (2 types of retainers and 2 types of bonding protocol)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bonding with rubberdam (Experimental): The retainer is bonded under rubber dam isolation
  Interventions: Device: Twistflex retainer; Device: Orthoflex retainer
- Bonding under relative isolation (Active Comparator): The retainer is bonded under relative isolation (hygrophormic suction, cotton pads)
  Interventions: Device: Twistflex retainer; Device: Orthoflex retainer

INTERVENTIONS:
Device: Twistflex retainer — twisted 0.0195 dead-soft coaxial wire (Respond; Ormco, Orange, Calif)
Device: Orthoflex retainer — Ortho-flextech (Reliance orthodontic products, Itasca III, USA)

SUMMARY:
Comparson of efficiency and effectiveness of twisted/coaxial and linked retainers, placed under relative versus absolute isolation.

DETAILED DESCRIPTION:
The domain of orthodontic retention is controversial. Orthodontic retention is the final step in an orthodontic procedure, and is performed after removal of the orthodontic appliance. Its goal is to prevent the relapse in occlusion or positioning of the teeth. Every patient will need some form of retention to maintain the ideal result. The bonded retainer is frequently used in the lower incisor region. It is capable to prevent relapse of orthodontic treatment but prevents tertiary crowding as well. Advantages of fixed retainers are in general no need for compliance and optimal aesthetics. The retention wire can stay in place for many years. Currently, there is a tendency towards lifelong retention. Disadvantages are more plaque and calculus accumulation, and possibly a poorer periodontal index.

Many types of bonded retainers with different properties could be bonded, each with different effects on periodontal health, potentially a different ability to maintain alignment, and different amounts of failure.

Different types of failure of fixed bonded retainers are possible. When the retainer does not stay in place and is debonded, this is is described as failure. It is also possible the retainer maintains bonded but shows unwanted tooth movement in the bonded teeth. This can also be described as a failure.

Bonding of the retention wire is a technique sensitive process. Correct and passive bonding could prevent debonding of the retainers. To eliminate moisture in the bonding process, it is possible to place a rubberdam before bonding the retainer.

One aim of this study is to compare two types of bonded retainer: the standard coaxial or twisted retainer. The other aim is to compare two bonding protocols with and without rubberdam isolation

Two general PICO questions can be formulated:

In an orthodontic patient (P), will fixed retention with a Ortho-flextech tm (Reliance orthodontic products, Itasca III, USA) (I) as compared to a 0.0195 in dead-soft coaxial wire (Respond; Ormco, Orange, Calif). (C) result in a more effective or efficient retention treatment (O)?

In an orthodontic patient (P), will placement of the retainer with rubber dam (I) result in less debonding (O) as compared to relative isolation with cotton rolls (C)?

Efficiency: is the procedure faster or cheaper than the alternative? Effectiveness: is the procedure better in maintaining the end result of treatment than the alternative? Are there less biomechanical or biological side effects?

ELIGIBILITY:
Inclusion Criteria:

* Fixed orthodontic appliances upper and lower jaw
* Patient stays for 2 years in Belgium
* Parents consent
* Proper oral hygiene

Exclusion Criteria:

* Orthognathic surgery
* Craniofacial disorders
* Cleft lip palate patients
* Orthodontic treatment without fixed appliances
* Extra retention other than bonded wire in the lower jaw

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Little Irregularity index | Measured before removing braces (T0), after 6 months (T1), 1 year (T2) and 2 years (T3)
  Stability of treatment. The index measures the distance, in millimetres, between the contact points of crooked teeth, and then adds them together. Therefore,the Irregularity Index is the sum of all the displaced contacts between the anterior teeth (canine to canine)

SECONDARY OUTCOMES:
Failure of the retainer (1) | Through study completion (2 years)
  Debonding of the retainer is registered, the date and place of reparation.
Failure of the retainer (2) | Through study completion (2 years)
  Possible activation (unwanted tooth movement possible torque differences) is checked after treatment.
Periodontal index- periodontal status | Measured before removing braces (T0), after 6 months (T1), 1 year (T2) and 2 years (T3)
  A periodontal status of the 6 anterior teeth is made, measuring probing depth 6 places per teeth
Periodontal index- BoP | Measured before removing braces (T0), after 6 months (T1), 1 year (T2) and 2 years (T3)
  Bleeding on probing is registered after the periodontal status (%)
Periodontal index- plaque | Measured before removing braces (T0), after 6 months (T1), 1 year (T2) and 2 years (T3)
  Plaque measurement (%)

CONTACTS AND LOCATIONS:
Overall Officials: Guy De Pauw, Prof, Study Chair — Head of orthodontics
Locations (1):
- University of Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stormann I, Ehmer U. A prospective randomized study of different retainer types. J Orofac Orthop. 2002 Jan;63(1):42-50. doi: 10.1007/s00056-002-0040-6. English, German. PMID 11974451
- [Background] Engeler OG, Dalstra M, Arnold DT, Steineck M, Verna C. In vitro comparison of the torsional load transfer of various commercially available stainless-steel wires used for fixed retainers in orthodontics. J Orthod. 2021 Jun;48(2):118-126. doi: 10.1177/1465312520972402. Epub 2020 Nov 24. PMID 33231109
- [Background] Ferreira LA, Sapata DM, Provenzano MGA, Hayacibara RM, Ramos AL. Periodontal parameters of two types of 3 x 3 orthodontic retainer: a longitudinal study. Dental Press J Orthod. 2019 Aug 1;24(3):64-70. doi: 10.1590/2177-6709.24.3.064-070.oar. PMID 31390451
- [Background] Sifakakis I, Eliades T, Bourauel C. Residual stress analysis of fixed retainer wires after in vitro loading: can mastication-induced stresses produce an unfavorable effect? Biomed Tech (Berl). 2015 Dec;60(6):617-22. doi: 10.1515/bmt-2015-0013. PMID 26057215
- [Background] Liebenberg WH. Extending the use of rubber dam isolation: alternative procedures. Part II. Quintessence Int. 1993 Jan;24(1):7-17. PMID 8511260
- [Background] Arnold DT, Dalstra M, Verna C. Torque resistance of different stainless steel wires commonly used for fixed retainers in orthodontics. J Orthod. 2016 Jun;43(2):121-9. doi: 10.1080/14653125.2016.1155814. Epub 2016 Apr 22. PMID 27104351
- [Background] Arnone R. Bonding orthodontic lower 3 to 3 retainers with a rubber dam: a second generation step-by-step procedure. Am J Orthod Dentofacial Orthop. 1999 Oct;116(4):432-4. doi: 10.1016/s0889-5406(99)70229-5. PMID 10511672
- [Background] Aldrees AM, Al-Mutairi TK, Hakami ZW, Al-Malki MM. Bonded orthodontic retainers: a comparison of initial bond strength of different wire-and-composite combinations. J Orofac Orthop. 2010 Jul;71(4):290-9. doi: 10.1007/s00056-010-9947-5. Epub 2010 Jul 30. English, German. PMID 20676816